CLINICAL TRIAL: NCT01498445
Title: An Open-Label, Phase I/II Study of Two Different Schedules of Dasatinib (Sprycel) and Decitabine (Dacogen) Used in Combination for Patients With Accelerated or Blastic Phase Chronic Myelogenous Leukemia (Protocol CA180357)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated early during the phase II portion of the study due to slow enrollment.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0333; CA180357 (Other: Bristol-Myers Squibb); NCI-2012-00014 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Leukemia
Keywords: Leukemia; Chronic myelogenous leukemia; Chronic myeloid leukemia; CML; Accelerated phase; Blastic phase; Dasatinib; BMS-354825; Sprycel; Decitabine; Dacogen
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Blast Crisis | interventions — Dasatinib; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase I - Dasatinib 100 mg + Decitabine 10 mg/m2 (Experimental): Less Intensive, Schedule A1 Dasatinib 100 mg daily by mouth ; Decitabine 10 mg/m^2 by vein over 1 hour daily for 10 days; 28 day cycle.
  Interventions: Drug: Dasatinib; Drug: Decitabine
- Phase I - Dasatinib 100 mg + Decitabine 20 mg/m2 (Experimental): More Intensive, Schedule A2: Dasatinib 100 mg daily by mouth ; Decitabine ose 20 mg/m^2 by vein over 1 hour daily for 10 days; 28 day cycle.
  Interventions: Drug: Dasatinib; Drug: Decitabine
- Phase I - Dasatinib 140 mg + Decitabine 10 mg/m2 (Experimental): Less Intensive, Schedule B1 Dasatinib 140 mg daily by mouth ; Decitabine 10 mg/m^2 by vein over 1 hour daily for 10 days; 28 day cycle.
  Interventions: Drug: Dasatinib; Drug: Decitabine
- Phase I - Dasatinib 140 mg + Decitabine 20 mg/m2 (Experimental): More Intensive, Schedule B2 Dasatinib 140 mg daily by mouth ; Decitabine 20 mg/m^2 by vein over 1 hour daily for 10 days; 28 day cycle.
  Interventions: Drug: Dasatinib; Drug: Decitabine
- Phase II - Dasatinib 140 mg + Decitabine 10 mg/m2 (Experimental): Less Intensive, Schedule B1 Dasatinib 140 mg daily by mouth; Decitabine e 10 mg/m^2 by vein over 1 hour daily for 10 days; 28 day cycle.
  Interventions: Drug: Dasatinib; Drug: Decitabine
- Phase II - Dasatinib 140 mg + Decitabine 20 mg/m2 (Experimental): More Intensive, Schedule B2 Dasatinib140 mg daily by mouth; Decitabine 20 mg/m^2 by vein over 1 hour daily for 10 days; 28 day cycle.
  Interventions: Drug: Dasatinib; Drug: Decitabine

INTERVENTIONS:
Drug: Dasatinib — Starting Dose: 100 mg by mouth once daily of a 28 day cycle.
  Other Names: BMS-354825; Sprycel
Drug: Decitabine — Starting Dose (less intensive group) Schedule A: 10 mg/m2 by vein daily for 10 days of a 28 day cycle.
  Other Names: Dacogen
  Arms: Phase I - Dasatinib 100 mg + Decitabine 10 mg/m2; Phase I - Dasatinib 140 mg + Decitabine 10 mg/m2; Phase II - Dasatinib 140 mg + Decitabine 10 mg/m2
Drug: Decitabine — Starting Dose (more intensive group) Schedule B: 20 mg/m2 by vein daily for 10 days of a 28 day cycle.
  Other Names: Dacogen
  Arms: Phase I - Dasatinib 100 mg + Decitabine 20 mg/m2; Phase I - Dasatinib 140 mg + Decitabine 20 mg/m2; Phase II - Dasatinib 140 mg + Decitabine 20 mg/m2

SUMMARY:
The goal of this clinical research study is to learn if combining Sprycel (dasatinib) and Dacogen (decitabine) can help to control Chronic Myeloid Leukemia (CML). The dose level of decitabine will also be studied.

Dasatinib is designed to block the protein that is responsible for chronic myeloid leukemia.

Decitabine is designed to affect the mechanism that cells use to control the expression of certain genes, some of which are important in the progression of CML.

This is an investigational study. Dasatinib is FDA approved and commercially available for the treatment of patients with certain types of CML.

Decitabine is FDA approved for the treatment of patients with myelodysplastic syndrome.

The combination of these drugs to treat CML is investigational.

Up to 84 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group and dose level based on when you join this study and the side effects that are seen. Your doctor will discuss this with you in more detail.

There will be up to 5 doses of dasatinib tested in Phase 1. The first 3 participants will receive a lower dose of therapy. If no major side effects are seen in these participants, the next participants will receive a higher dose. Once a dose is identified that is well-tolerated for most participants, that dose will be used for all new participants. If you are in Phase 2, you will receive a dose level tested in Phase 1.

You will receive one of 2 doses of decitabine. What dose you receive is determined by chance (like a coin toss).

Study Administration:

Each cycle is 28 days.

You will take dasatinib by mouth 1 time a day.

You will receive decitabine by vein for 10 days of each cycle. If the doctor thinks it is in your best interest, you may receive decitabine for fewer days each cycle (5 days instead of 10 days). Your doctor will decide how many doses you will take based on side effects you may have and the status of the disease.

If you have severe side effects from the study drug, the study doctor may decide to stop drug dosing until your side effects improve.

You will be asked to keep a study diary that will be reviewed at scheduled study visits. In the diary, you will record when you take the study drug.

Study Visits:

At every visit, you will be asked about any side effects you may have had and to list any drugs you may be taking.

Every week for the first 3 cycles and then every 2-4 weeks after that, blood (about 1 tablespoon) will be drawn to check your blood cell counts.

About 1 week after your first dose, you will have an ECG.

Every 1-2 weeks for the first 3 cycles and then every 4-8 weeks after that, blood (about 1 tablespoon) will be drawn to test your kidney and liver function.

Every 1-3 months, blood (about 1 tablespoon) will be drawn for genetic testing.

Before the start of Cycle 2, every 2-4 cycles after that for the first year, and then every 6 cycles after that, you will have a complete physical exam.

Before the start of Cycle 2, every 3 cycles after that during the first year, then every 4-6 cycles (as needed) you will have a bone marrow aspirate to check the status of the disease.

After Cycle 6, the number of blood draws and bone marrow collections may be changed.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 years of age or older with CML-AP, CML-BP or Philadelphia chromosome-positive acute myeloid leukemia defined as follows: CML-AP is defined by the presence of 15-29% blasts in peripheral blood (PB) or bone marrow (BM), >/= 20% basophils in PB or BM, >/= 30% blasts plus promyelocytes (with blasts <30%) in PB or BM, <100 x10(9)/L platelets unrelated to therapy, or by clonal cytogenetics evolution (i.e., the presence of cytogenetic abnormalities other than the Philadelphia chromosome); CML-BP is defined by the presence of >/= 30% blasts in the bone marrow and/or peripheral blood or the presence of extramedullary disease.
2. Patients are eligible whether they have received or not prior TKI therapy. For the phase I portion of the study, patients who had received prior therapy with dasatinib should have been able to tolerate the dose equivalent to the starting dose of dasatinib in the dose level at which the patient is being entered. Patients who previously received dasatinib but never at the dose being proposed are eligible provided they tolerated the maximum dose they were prescribed with no grade 3-4 toxicity not responding to optimal management.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-3.
4. Men and women of childbearing potential should practice 2 methods of contraception; 1 method must be highly effective and a second method must be either highly effective or less effective. Men and women of childbearing potential are defined as: a male that has not been surgically sterilized or a female that has not been amenorrheic for at least 12 consecutive months or that has not been surgically sterilized. Patients must use birth control during the study and for 3 months after the last dose of study drug if they are sexually active.
5. Women of childbearing potential must have a pregnancy test at screening.
6. Signed informed consent.
7. Patients must have been off all prior therapy for CML for 2 weeks prior to start of study therapy and recovered from the toxic effects of that therapy. Exceptions to these are hydroxyurea and Tyrosine kinase inhibitor (TKIs) (including but not limited to imatinib, nilotinib, and bosutinib) which should be discontinued >/= 24 hrs prior to the start of therapy. Patients who are receiving dasatinib prior to enrollment do not have to discontinue this agent prior to start of study therapy.
8. Adequate organ function: Serum creatinine </= 2.0 mg/dl or creatinine clearance >/=60 mL/min; Total bilirubin </= 1.5 x upper limit of normal (ULN) (unless considered due to Gilbert's syndrome or hemolysis); Alanine aminotransferase (ALT) </= 3 x ULN unless considered due to leukemic involvement.

Exclusion Criteria:

1. New York Heart Association (NYHA) cardiac class 3-4 heart disease.
2. Cardiac disease including: Uncontrolled angina within 3 months. Diagnosed or suspected congenital long QT syndrome; Any history of clinically significant ventricular arrhythmias (eg, ventricular tachycardia, ventricular fibrillation, or Torsades de pointes); Prolonged QTc interval on pre-entry electrocardiogram (> 470 msec) on the Fridericia's correction; Uncontrolled hypertension (defined for this protocol as sustained systolic BP >/=150 and diastolic >/=100); Patients currently taking drugs that are generally accepted to have a risk of causing Torsades de Pointes.
3. Serious uncontrolled medical disorder or uncontrolled active systemic infection or current unstable or decompensated respiratory or cardiac conditions which makes it undesirable or unsafe for the patient to participate in the study.
4. Patients with known, clinically significant pericardial or pleural effusion.
5. History of significant bleeding disorder unrelated to cancer, including diagnosed congenital bleeding disorders (e.g., von Willebrand's disease), or diagnosed acquired bleeding disorders within one year (e.g., acquired anti-factor VIII antibodies).
6. Subject is receiving potent inhibitors of CYP3A4; for such medications, a wash-out period of >/= 7 days is required prior to starting dasatinib unless discontinuation or substitution of such an inhibitor is not in the best interest of the patient as determined by the investigator. These include the following medications: itraconazole, ketoconazole, miconazole, voriconazole; amprenavir, atazanavir, fosamprenavir, indinavir, nelfinavir, ritonavir; ciprofloxacin, clarithromycin, diclofenac, doxycycline, enoxacin, isoniazid, ketamine, nefazodone, nicardipine, propofol, quinidine, telithromycin. In instances where use of these agents is felt to be required for the best management of the patients, inclusion of such a patients should be discussed with PI and the rationale documented.
7. Females who are pregnant or are currently breastfeeding.
8. Patients that are eligible (including having available donor) and willing to receive an allogeneic stem cell transplant within 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-06-12 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: June 2012 to April 2018
Groups:
- Phase I Schedule A1: Dasatinib 100mg + Decitabine 10 mg/m2
- Phase I Schedule A2: Dasatinib 100 mg + Decitabine 20 mg/m2
- Phase I Schedule B1; Phase II B1: Dasatinib 140 mg + Decitabine 10 mg/m2
- Phase I Schedule B2: Dasatinib 140 mg+ Decitabine 20 mg/m2
- Phase II B2: Dasatinib 140 mg + Decitabine 20 mg/m2
Period: Overall Study
Arm/Group | Phase I Schedule A1 | Phase I Schedule A2 | Phase I Schedule B1 | Phase I Schedule B2 | Phase II B1 | Phase II B2
Started | 4 | 3 | 8 | 8 | 4 | 5
Completed | 4 | 3 | 7 | 6 | 3 | 4
Not Completed | 0 | 0 | 1 | 2 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Screen Failure | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase I - Dasatinib 100 mg + Decitabine 10 mg/m2: Less Intensive, Schedule A1 Dasatinib starting dose of 100 mg by mouth daily; Decitabine starting dose 10 mg/m2 by vein over 1 hour daily for 10 days; 28 day cycle.
  Dasatinib: Starting Dose: 100 mg by mouth once daily of a 28 day cycle.
  Decitabine: Starting Dose (less intensive group) Schedule A: 10 mg/m2 by vein daily for 10 days of a 28 day cycle.
- Phase I - Dasatinib 100 mg + Decitabine 20 mg/m2: More Intensive, Schedule A2: Dasatinib starting dose 100 mg by mouth daily; Decitabine starting dose 20 mg/m2 by vein over 1 hour daily for 10 days; 28 day cycle.
  Dasatinib: Starting Dose: 100 mg by mouth once daily of a 28 day cycle.
  Decitabine: Starting Dose (more intensive group) Schedule B: 20 mg/m2 by vein daily for 10 days of a 28 day cycle.
- Phase I - Dasatinib 140 mg + Decitabine 10 mg/m2; Phase II - Dasatinib 140 mg + Decitabine 10 mg/m2: Less Intensive, Schedule B1 Dasatinib starting dose of 140 mg by mouth daily; Decitabine starting dose 10 mg/m2 by vein over 1 hour daily for 10 days; 28 day cycle.
  Dasatinib: Starting Dose: 100 mg by mouth once daily of a 28 day cycle.
  Decitabine: Starting Dose (less intensive group) Schedule A: 10 mg/m2 by vein daily for 10 days of a 28 day cycle.
- Phase I - Dasatinib 140 mg + Decitabine 20 mg/m2; Phase II - Dasatinib 140 mg + Decitabine 20 mg/m2: More Intensive, Schedule B2 Dasatinib starting dose of 140 mg by mouth daily; Decitabine starting dose 20 mg/m2 by vein over 1 hour daily for 10 days; 28 day cycle.
  Dasatinib: Starting Dose: 100 mg by mouth once daily of a 28 day cycle.
  Decitabine: Starting Dose (more intensive group) Schedule B: 20 mg/m2 by vein daily for 10 days of a 28 day cycle.
- Total: Total of all reporting groups
Arm/Group | Phase I - Dasatinib 100 mg + Decitabine 10 mg/m2 | Phase I - Dasatinib 100 mg + Decitabine 20 mg/m2 | Phase I - Dasatinib 140 mg + Decitabine 10 mg/m2 | Phase I - Dasatinib 140 mg + Decitabine 20 mg/m2 | Phase II - Dasatinib 140 mg + Decitabine 10 mg/m2 | Phase II - Dasatinib 140 mg + Decitabine 20 mg/m2 | Total
Number analyzed (Participants) | 4 | 3 | 8 | 8 | 4 | 5 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7 | 7 | 4 | 2 | 27
  >=65 years | 0 | 0 | 1 | 1 | 0 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 2 | 2 | 1 | 12
  Male | 3 | 0 | 5 | 6 | 2 | 4 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3 | 1 | 0 | 7
  White | 3 | 3 | 6 | 4 | 1 | 5 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 8 | 8 | 4 | 5 | 32

OUTCOME MEASURES:

1. Primary Outcome: Ph I Study: Maximum Tolerated Dose (MTD) Dasatinib
Description: Maximum tolerated dose (MTD) defined as highest dose at which 0 of 3 or </= 1/6 participant experience a first cycle dose limiting toxicity (DLT).
Time Frame: End of first 28-day cycle
Population: Participants who did not complete 2 cycles of therapy were ineligible for response. Maximum Tolerate Dose (MTD) was not done for the Phase II portion of the study, therefore zero participants in the Phase II arms were analyzed for this outcome.
Measure: Number; unit: Milligrams
Arm/Group | Phase I - Dasatinib 100 mg + Decitabine 10 mg/m2 | Phase I - Dasatinib 100 mg + Decitabine 20 mg/m2 | Phase I - Dasatinib 140 mg + Decitabine 10 mg/m2 | Phase I - Dasatinib 140 mg + Decitabine 20 mg/m2 | Phase II - Dasatinib 140 mg + Decitabine 10 mg/m2 | Phase II - Dasatinib 140 mg + Decitabine 20 mg/m2
Number analyzed (Participants) | 4 | 3 | 7 | 6 | 0 | 0
Milligrams | NA — There were no dose limiting toxicities for this treatment arm | NA — There were no dose limiting toxicities for this treatment arm | 140 | 140 |  |

2. Secondary Outcome: Number of Participants With Hematologic Responses During First 3 Months of Treatment
Description: Number of participants with hematologic response (HR) to therapy during first 3 months of combination dasatinib and decitabine therapy, where HR defined as any hematologic response observed during the first 3 months of treatment. Overall Hematologic Response (OHR) is defined as complete hematologic response (CHR), no evidence of leukemia (NEL) or minor hematologic response (MiHR)
Time Frame: 3 months
Population: 1 participant in Ph 1 Dasatinib 140 mg + Decitabine 10 mg/m^2 arm was not evaluable for response. 2 participants in the Ph 1 Dasatinib 140 mg + Decitabine 20 mg/m^2 arm were not evaluable for response. 1 participant in Ph II Dasatinib 140 mg + Decitabine 10mg/m^2 and 1 participant in Ph II Dasatinib 140 mg + Decitabine 20mg/m^2 failed screening.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Dasatinib 100 mg + Decitabine 10 mg/m2 | Phase I - Dasatinib 100 mg + Decitabine 20 mg/m2 | Phase I - Dasatinib 140 mg + Decitabine 10 mg/m2 | Phase I - Dasatinib 140 mg + Decitabine 20 mg/m2 | Phase II - Dasatinib 140 mg + Decitabine 10 mg/m2 | Phase II - Dasatinib 140 mg + Decitabine 20 mg/m2
Number analyzed (Participants) | 4 | 3 | 7 | 6 | 3 | 4
Participants | 3 | 1 | 5 | 4 | 3 | 3

3. Secondary Outcome: Overall Survival
Description: Overall Survival will be measured from the date treatment is started to the date of death or last follow-up.
Time Frame: Up to seven years
Population: 1 participant in Ph 1 Dasatinib 140 mg + Decitabine 10 mg/m^2 arm was not evaluable for response. Two participants in the Ph 1 Dasatinib 140 mg + Decitabine 20 mg/m^2 arm were not evaluable for response.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I - Dasatinib 100 mg + Decitabine 10 mg/m2 | Phase I - Dasatinib 100 mg + Decitabine 20 mg/m2 | Phase I - Dasatinib 140 mg + Decitabine 10 mg/m2 | Phase I - Dasatinib 140 mg + Decitabine 20 mg/m2 | Phase II - Dasatinib 140 mg + Decitabine 10 mg/m2 | Phase II - Dasatinib 140 mg + Decitabine 20 mg/m2
Number analyzed (Participants) | 4 | 3 | 7 | 6 | 3 | 4
Months | 12.0 [0.6 to 36.8] | 7.0 [2.3 to 82.8] | 57.8 [0.9 to 79.4] | 58.2 [3.6 to 58.2] | 62.0 [6.0 to 62.0] | 37.5 [9.6 to 37.5]

4. Secondary Outcome: Duration of Response
Description: Duration of Response will be measured from the date the given response is achieved to the date the response is first known to be lost
Time Frame: up to seven years
Population: as for outcome 3
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I - Dasatinib 100 mg + Decitabine 10 mg/m2 | Phase I - Dasatinib 100 mg + Decitabine 20 mg/m2 | Phase I - Dasatinib 140 mg + Decitabine 10 mg/m2 | Phase I - Dasatinib 140 mg + Decitabine 20 mg/m2 | Phase II - Dasatinib 140 mg + Decitabine 10 mg/m2 | Phase II - Dasatinib 140 mg + Decitabine 20 mg/m2
Number analyzed (Participants) | 4 | 3 | 7 | 6 | 3 | 4
Months | 36.8 [1.2 to 36.8] | 82 [82 to 82] | 57.8 [.09 to 79.4] | 58 [37 to 58] | 61 [1.5 to 61.0] | 37 [30 to 37]

ADVERSE EVENTS:
Time Frame: Up to seven years
Arm/Group | Phase I - Dasatinib 100 mg + Decitabine 10 mg/m2 | Phase I - Dasatinib 100 mg + Decitabine 20 mg/m2 | Phase I - Dasatinib 140 mg + Decitabine 10 mg/m2 | Phase I - Dasatinib 140 mg + Decitabine 20 mg/m2 | Phase II - Dasatinib 140 mg + Decitabine 10 mg/m2 | Phase II - Dasatinib 140 mg + Decitabine 20 mg/m2
All-Cause Mortality (participants affected / at risk) | 1/4 | 1/3 | 2/8 | 0/8 | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 3/4 | 3/3 | 7/8 | 6/8 | 3/4 | 4/5
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 7/8 | 8/8 | 3/4 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Dasatinib 100 mg + Decitabine 10 mg/m2 (N=4) | Phase I - Dasatinib 100 mg + Decitabine 20 mg/m2 (N=3) | Phase I - Dasatinib 140 mg + Decitabine 10 mg/m2 (N=8) | Phase I - Dasatinib 140 mg + Decitabine 20 mg/m2 (N=8) | Phase II - Dasatinib 140 mg + Decitabine 10 mg/m2 (N=4) | Phase II - Dasatinib 140 mg + Decitabine 20 mg/m2 (N=5)
Abdominal Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenic Fever (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Fever (General disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Gastric Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General Administration Site (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 2 (6) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital Edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal and Urinary Disorders (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Respiratory Thoracic and Mediastinal Disorders Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic Event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Dasatinib 100 mg + Decitabine 10 mg/m2 (N=4) | Phase I - Dasatinib 100 mg + Decitabine 20 mg/m2 (N=3) | Phase I - Dasatinib 140 mg + Decitabine 10 mg/m2 (N=8) | Phase I - Dasatinib 140 mg + Decitabine 20 mg/m2 (N=8) | Phase II - Dasatinib 140 mg + Decitabine 10 mg/m2 (N=4) | Phase II - Dasatinib 140 mg + Decitabine 20 mg/m2 (N=5)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema (General disorders) | 1 (1) | 1 (2) | 3 (3) | 2 (3) | 2 (2) | 0 (0)
Elevated Amylase (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated Lipase (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 5 (6) | 2 (2) | 1 (1)
Hyperbilirubinemia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 5 (6) | 2 (3) | 3 (4)
Mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 4 (5) | 3 (4) | 2 (2) | 0 (0)
Neutropenia (Investigations) | 0 (0) | 0 (0) | 1 (2) | 4 (5) | 1 (3) | 2 (2)
Neutropenic Fever (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (9) | 0 (0) | 4 (4) | 3 (8) | 1 (3) | 2 (6)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (6) | 1 (1) | 2 (3)
Hemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (5) | 1 (2) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Weight Gain (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot Flashes (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT01498445/Prot_SAP_000.pdf